CLINICAL TRIAL: NCT03671499
Title: A Pilot Study for Testing the Feasibility and Efficacy of Text Messaging and Newsletter as a Strategy for Interrupting Sedentary Behavior (Sit Less, Move More)
Brief Title: A Study for Testing Text Messaging and Newsletter as a Strategy for Interrupting Sedentary Behavior
Acronym: SLMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Consortium of Multiple Sclerosis Centers (Other)
Responsible Party: Principal Investigator, Robert W Motl, Primary Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0000518843
Record Dates: First submitted 2018-09-10; First posted 2018-09-14 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis
Keywords: sedentary behavior; physical activity
MeSH Terms: conditions — Multiple Sclerosis; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social Cognitive Theory based text messages (Experimental): The study only contains 1 arm. All participants will receive the same experimental protocol. Participants will receive daily text messages and bi-weekly newsletters for reducing sedentary behavior based on Social Cognitive Theory.
  Interventions: Behavioral: Social Cognitive Theory based text messages

INTERVENTIONS:
Behavioral: Social Cognitive Theory based text messages — Participants receive daily text messages and bi-weekly newsletters with information about reducing sitting behavior and increasing physical activity.

SUMMARY:
The study will examine the possibility of reducing sedentary behavior (SB) in African Americans with MS. SB consists of any waking activities that are done lying or sitting and do not demand significant physical effort (e.g., watching television, using the computer). SB is a major public health issue because it is associated with mortality and higher probabilities of presenting with health conditions and morbidity. There is indication that SB is related to physical disability, which is the inability of performing daily activities independently. This outcome is of high concern for persons with MS, especially those from underserved groups, such as African Americans. Thus, reducing the amount of time that people with MS spend in SB is important, but it is hard to find ways of doing so in large groups of people with MS. One possibility is to use text-messages to inform people about the necessity and benefits of interrupting SB by standing up, walking, or doing another activity. Text-messages are an ideal way to prompt behavior change because almost everyone owns a cellphone/smartphone in today's world. Considering this potential, the investigators will be studying whether or not it is possible to have a small group of African Americans with MS spend less time in SB by sending informative text-messages prompting individuals to stand-up and move around. This study will be used to inform the development of a much larger study that will aim to reduce SB in a very large sample of persons with MS.

DETAILED DESCRIPTION:
The investigators are conducting a pilot study to examine the feasibility and efficacy of a technology-based behavior change intervention for reducing SB in African Americans with MS located in the United States. The intervention combines text message- and print-based approaches for behavior change based on Social Cognitive Theory (SCT). SCT-based content will be the active component for changing SB, while cellphone text messages and print newsletter will be the delivery mechanism. The use of cellphone to deliver the intervention content is based, in part, on the fact that cellphone is an ordinary form of communication in today's world, providing an optimal medium for reaching large groups of people remotely. The study will yield major advancement in identifying the feasibility and efficacy of interrupting and reducing SB via a technology-based intervention in African Americans with MS, a segment of the MS population that has been underrepresented in MS therapeutic management studies. If successful, this research will lay the foundation for applying the current strategy in large-scale interventions including African Americans and possibly other minority groups with MS.

The intervention will be 12 weeks and divided into two parts. Part 1: Weeks 1-6 will focus on interrupting long periods of SB. At the beginning of the first week, participants will receive a packet containing print material providing lay information on what constitutes SB and examples of such behavior, highlighting the importance of interrupting prolonged periods of SB and the associated health benefits. The aim of the packet is to provide the basis to introduce the key element (i.e., SCT-based instructional cellphone text-messages) of the intervention. This will occur during the following six weeks, wherein participants will receive two text-messages/day (i.e., morning and afternoon) on the importance and health benefits of interrupting SB hourly. The text-messages will prompt individuals to interrupt SB by standing still, standing while performing tasks, or walking around. The text-messages will include further tips and strategies for interrupting SB. The investigators have previously developed a computerized messaging system that will be used to send the text-messages twice a day in the proposed intervention. The investigators will supplement the text messaging by sending bi-weekly SCT-based newsletters to participants that highlight ways of overcoming difficulties in effectively interrupting SB. The SCT content for the messages and newsletter has been created in previous research and will be revised for the proposed intervention. Part 2: Weeks 7-12 will focus on replacing SB with light PA. On the first day of week 7, participants will receive a second packet of print material explaining the concept of light PA and emphasizing the importance of moving more daily. The print material will highlight the benefits of replacing SB with light PA and will contain instructions for goal setting (i.e., target number of steps/day) and self-monitoring of daily PA, including receive a pedometer and a log for recording total steps/day. Similar to part 1, the key element for intervention delivery will be the SCT-based instructional cellphone text-messages, which participants will receive during the second six-week intervention period. More specifically, they will receive two text-messages/day on the importance and health benefits of replacing SB with light PA. The text-messages will recommend participants to watch for prolonged periods of SB and try and substitute these for light PA, such as light intensity walking and light-intensity focal exercise (e.g., stationary walk, marching). The text-messages will also remind participants to use the pedometer to set incremental personal goals for steps/day and to gauge the replacement of SB with light PA by watching the pedometer readings. The investigators further will include tips and strategies for replacing SB with light PA based on common daily activities. Bi-weekly SCT-based newsletters will be used to supplement the stimulus from the text-messages, by reinforcing the importance of sitting less and moving more.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Definite diagnosis of MS
* Relapse free in the last 30 days
* Ambulatory with or without assistance
* Having a Patient-Determined Disease Steps score of 0-5
* Daily engagement in sedentary behavior ≥ 480 min/day
* Health contribution score of <14 calculated from the Godin Leisure-Time Exercise Questionnaire
* Absence of major musculoskeletal problems, and/or cardiovascular, cardiopulmonary, and/or metabolic diseases that can influence physical activity and sedentary behavior levels

Exclusion Criteria:

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Change in sedentary behavior evaluated with activity monitors | Assessments will be conducted at baseline and at the midpoint of the experiment (intervention week 6)
  Activity monitors are Actigraph accelerometers that participants will wear on an elastic belt around their waist for 7 days. These activity monitors measure how frequently and how much an individual moves.
Change in sedentary behavior evaluated with activity monitors | Assessments will be conducted at the midpoint of the intervention (intervention week 6) and at at the end of the intervention (immediately after intervention week 12).
  Activity monitors are Actigraph accelerometers that participants will wear on an elastic belt around their waist for 7 days. These activity monitors measure how frequently and how much an individual moves.
Change in sedentary behavior evaluated with activity monitors | Assessments will be conducted at baseline and at at the end of the intervention (immediately after intervention week 12).
  Activity monitors are Actigraph accelerometers that participants will wear on an elastic belt around their waist for 7 days. These activity monitors measure how frequently and how much an individual moves.
Change in physical activity evaluated with activity monitors | Assessments will be conducted at baseline and at the midpoint of the experiment (intervention week 6)
  Activity monitors are Actigraph accelerometers that participants will wear on an elastic belt around their waist for 7 days. These activity monitors measure how frequently and how much an individual moves.
Change in physical activity evaluated with activity monitors | Assessments will be conducted at the midpoint of the intervention (intervention week 6) and at at the end of the intervention (immediately after intervention week 12).
  Activity monitors are Actigraph accelerometers that participants will wear on an elastic belt around their waist for 7 days. These activity monitors measure how frequently and how much an individual moves.
Change in physical activity evaluated with activity monitors | Assessments will be conducted at baseline and at at the end of the intervention (immediately after intervention week 12).
  Activity monitors are Actigraph accelerometers that participants will wear on an elastic belt around their waist for 7 days. These activity monitors measure how frequently and how much an individual moves.

SECONDARY OUTCOMES:
Quality of Life will be evaluated with the 36-Item Short Form Health Survey (SF-36 questionnaire). | Assessments will be conducted at baseline and at the midpoint of the experiment (intervention week 6)
  The SF-36 questionnaire is a 36 item self-report questionnaire designed to assess patient health status. The questionnaire is scored on 8 sections: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Scores are transformed into a 0-100 scale with 0 equivalent to maximum disability and 100 equivalent to no disability.
Quality of Life will be evaluated with the 36-Item Short Form Health Survey (SF-36 questionnaire). | Assessments will be conducted at the midpoint of the intervention (intervention week 6) and at at the end of the intervention (immediately after intervention week 12).
  The SF-36 questionnaire is a 36 item self-report questionnaire designed to assess patient health status. The questionnaire is scored on 8 sections: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Scores are transformed into a 0-100 scale with 0 equivalent to maximum disability and 100 equivalent to no disability.
Quality of Life will be evaluated with the 36-Item Short Form Health Survey (SF-36 questionnaire). | Assessments will be conducted at baseline and at at the end of the intervention (immediately after intervention week 12).
  The SF-36 questionnaire is a 36 item self-report questionnaire designed to assess patient health status. The questionnaire is scored on 8 sections: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Scores are transformed into a 0-100 scale with 0 equivalent to maximum disability and 100 equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Motl, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Baird JF, Sasaki JE, Sandroff BM, Cutter G, Motl RW. An Intervention for Changing Sedentary Behavior Among African Americans With Multiple Sclerosis: Protocol. JMIR Res Protoc. 2019 May 1;8(5):e12973. doi: 10.2196/12973. PMID 31042149